CLINICAL TRIAL: NCT04722614
Title: The Effect of Music and Essential Oil on Agitation in Mechanically Ventilated Patients
Brief Title: Music and Essential Oil in Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1112021
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2021-01

CONDITIONS: Agitation
Keywords: Mechanical ventilation; Music therapy; Essential oil; Bergamot oil
MeSH Terms: conditions — Psychomotor Agitation | interventions — Music Therapy; Oils, Volatile

STUDY DESIGN:
Intervention Model Description: Three-group pre-test and repeated post-test study
Who Masked: Care Provider
Masking Description: Computer generated randomization (www.randomizer.org) will be used to randomly assign patients to groups. Information of allocation was available to the principal researcher only. Patients will be assigned in sequential numbers that will be placed in an opaque, sealed envelope by the researcher. After patients enrollment, the envelope will be opened. The nurses could not be blinded to the allocation because of the nature of the intervention. However, the outcome assessment of the patients was blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Mechanically ventilated patients who will be subjected to the routine unit intervention for agitation
  Interventions: Other: Control
- Music group (Experimental): Mechanically ventilated patients who will listen to classic music
  Interventions: Other: Music
- Essential oil group (Experimental): Mechanically ventilated patients who will inhale bergamot oil
  Interventions: Other: Essential oil

INTERVENTIONS:
Other: Music — Classic music hearing at amplitude approximately 60-80 dB using MP3 player connected to headphone with noise canceling property
  Arms: Music group
Other: Essential oil — Bergamot oil inhalation through a piece of cotton gauze (2 × 2 cm square shape) with 0.5 cc of bergamot oil. It will be attached to the collar of the patient's clothes gown, approximately 15 cm below their nose.
  Arms: Essential oil group
Other: Control — The routine intensive care unit sedation protocol
  Arms: Control group

SUMMARY:
The study aims to assess the effect of using music and essential oil on agitation in mechanically ventilated patients. Listening to classical relaxation music, and inhalation to bergamot oil will be used in this study.

DETAILED DESCRIPTION:
Agitation in critically ill patients is a phenomenon that can compromise patient safety and assistance during intensive care unit (ICU) hospitalizations. This trial will be conducted in five general intensive care unit. One hundred and twenty patients will be enrolled in this study divided into three equal groups (40 patients in each group). Group A is the control group. Group B is music group. Group C is essential oil group. Agitated mechanically ventilated patients will be randomly assigned to one of the three groups. Each group will be subjected to its specific intervention and they will be monitored for seven days. Agitation score and frequency outcome will be assessed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Agitation with RASS score +2 or more
* Mechanical ventilation
* Patients with GCS 13-15

Exclusion Criteria:

* Psychiatric illness
* Cognitive disorders
* Neurological disorder
* Hearing deficit
* Smelling deficit
* Respiratory asthma
* Allergic rhinitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2021-04-11 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Agitation score | 7 days
  Agitation score is assessed by Richmond Agitation-Sedation Scale (RASS). The RASS is a 10-point scale ranging from -5 to +4. Levels from -1 to -5 denote increasing levels of sedation. Levels from +1 to +4 describe increasing levels of agitation. Zero score is the best response for the patient which is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: E A Hassan, Principal Investigator — Alexandria University
Locations (2):
- Egypt (2):
  - Alexandria Main University Hospital, Alexandria
  - Faculty of nursing, Alexandria

IPD SHARING:
Plan to Share IPD: No
Researchers are waiting to get approval from research committee to make individual participant data (IPD) available to other researchers